CLINICAL TRIAL: NCT06125119
Title: Development of Minimally Invasive Methodology for Diabetyping to Personalise Treatment to Realise Remission and Reversal of Type 2 Diabetes
Acronym: 2DIAREM
Status: Recruiting | Type: Observational
Sponsor: TNO (Other)
Responsible Party: Sponsor
Other Study IDs: NL83666.028.23
Record Dates: First submitted 2023-09-21; First posted 2023-11-09 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Lifestyle changes in diet and exercise can reverse type 2 diabetes (T2D), also referred to as T2D remission. Although combined lifestyle interventions for T2D remission are promising, not all persons react similarly to such 'one-size-fits-all' interventions. Research has shown that as a result of differences in T2D pathophysiology between individuals, different subgroups of T2D can be identified, that differ in which diet is most beneficial in the recovery of pancreatic beta-cell function. TNO and partners work on the development of the Diabetyping Lifestyle Intervention (DLI) for T2D subtypes that tailors the combined lifestyle intervention based on organ dysfunction (liver, muscle and/or pancreatic beta cell function) by using the Oral Glucose Tolerance Test (OGTT). Current diabetyping is invasive, needs to take place in a clinical setting, and therefore is not suited for scaling to application in the large T2D population of more than 1 million people. Therefore, less invasive, scalable alternatives are warranted.

Objective: The main objective of the 2DIAREM study is to develop minimally invasive alternatives of diabetyping. Two alternative sampling methods will be evaluated, finger pricks and continuous glucose monitoring (CGM). Data collected through these technologies may be used to predict OGTT indices and diabetypes to guide personalized lifestyle interventions for T2D patients. Furthermore, the investigators aim to develop and evaluate the minimally invasive diabetyping technology with algorithms based on finger prick sampling and multi-day CGM upon a standardized snack or multi-day CGM only under real-world conditions.

Study design: The study will be an observational study, lasting 20 days and consisting of three mornings with measurements.

Study population: A heterogenous group of people with overweight/(pre)diabetes type 2. The investigators aim for equal distribution among overweight/prediabetes, mild diabetes, and severe diabetes in the study population.

Intervention (if applicable): During the 20 days of monitoring participants are asked to undergo one OGTT and consume two times a standardized snack (Snelle Jelle (naturel 65 gram)) after an overnight fast. In between participants are asked to follow their usual lifestyle.

Main study parameters/endpoints: Continuously measured subcutaneous glucose, as well as, glucose and insulin, and c-peptide collected via capillary sampling for the development of algorithms predicting the different diabetypes and the underlying indices based on venous blood glucose and insulin.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The burden of this study consists of the application and removal of the continuous glucose monitor device, and the consumption of a sweet beverage (OGTT) and two standardized snacks and undergoing several capillary blood draws. The risks associated with participation can be considered negligible, and are mainly associated with the glucose sensor and the OGTT. The glucose sensor provides a small risk of adverse events including skin irritation, skin infection, and skin colouring. The OGTT poses a small risk of hypo- or hyperglycaemia and can lead to nausea. However, experienced medical professionals are present at the clinic and will closely monitor well-being and health status of the study participants. Benefits include that data collected through the technologies may be used to predict OGTT indices and diabetypes much less invasively and scalable to guide personalized lifestyle interventions for T2D patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with (pre)diabetes type 2;

  * BMI ≥27 kg/m2, including a heterogenous group of people/with overweight/prediabetes (without glucose lowering medication), and/or type 2 diabetes with or without glucose lowering medication.
* Aged 40 years or older
* Able and willing to sign the informed consent form
* Willing to comply with all study procedures

Exclusion Criteria:

* Type 1 diabetes
* Latent Autoimmune Diabetes (LADA)
* Skin allergy, eczema or known sensitivity for adhesives
* History of bariatric weight loss surgery
* Planned (bariatric) surgery during the 3 weeks monitoring period with the CGM
* Active cancer or chemotherapy or radiation within 2 years prior to participation
* A condition that would need an MRI during the 3 weeks monitoring period with the CGM
* Planned holiday during the 3 week GCM monitoring period
* (Night)shiftworkers
* Pregnancy and lactation
* Chronic medical condition, treatment, or medication other than diabetes that may affect glucose metabolism (HIV diagnosis, use of steroids or immunosuppressive drugs, etc.)
* 4 or more alcoholic drinks per day on a regular basis or use of recreational drugs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of people with overweight/prediabetes, mild diabetes and severe diabetes, as diagnosed by BMI, disease duration, medication use and CVD history. The three subpopulations are selected to ensure representative variability in OGTT response and diabetes subtypes.
Sampling Method: Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Glucose values (mmol/l) | In-study at day 3 and day 17 (venous and capillary) during 20 days with CGM
  Measured in venous blood, capillary blood and interstitial fluid (via the CGM) before and during the OGTT
Insulin (mIU/l) | In-study at day 3 and day 17 (venous and capillary)
  Measured in venous blood and capillary blood before and during the OGTT
c-peptide (nmol/l) | In-study at day 3 and day 17 (venous and capillary)
  Measured in venous blood and capillary blood before and during the OGTT
Diabetyping | End of study (after 20 days)
  Development of algorithms predicting the different diabetypes and the underlying indices with minimally invasive data collection (e.g. capillary blood sampling with sample tube/dry blood spot and CGM)

SECONDARY OUTCOMES:
Glucose values (mmol/l) | In-study at day 8 (capillary) and day 17 (venous and capillary) during 20 days with CGM
  Measured in capillary blood, venous and interstitial fluid (via the CGM) before and during the standardized snack
Insulin (mIU/l) | In-study at day 8 (capillary) and day 17 (venous and capillary)
  Measured in capillary blood, venous and interstitial fluid (via the CGM) before and during the standardized snack
c-peptide (nmol/l) | In-study at day 8 (capillary) and day 17 (venous and capillary)
  Measured in capillary blood, venous and interstitial fluid (via the CGM) before and during the standardized snack
Diabetyping | End of study (after 20 days)
  Assess the agreement between diabetyping based on a standardized snack as compared to the OGTT

OTHER OUTCOMES:
Self-reported experiences with capillary blood sampling in an at home setting | End of study (day 19)
  Via a self composed questionnaire with open and closed questions

CONTACTS AND LOCATIONS:
Locations (1):
- Reinier Haga, Leiden, Netherlands